CLINICAL TRIAL: NCT06296147
Title: A Randomized, Controlled Trial: Impact on Patient Experience in Patients Assigned to Virtual Reality Headset; Aromatherapy Patch; Virtual Reality + Aromatherapy; or Standard of Care for Transperineal Prostate Biopsy
Brief Title: Virtual Reality Headset and/or Aromatherapy for Patients Undergoing a Transperineal Prostate Biopsy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Responsible Party: Principal Investigator, Bruce Jacobs, Assistant Professor, University of Pittsburgh School of Medicine, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY23080006
Record Dates: First submitted 2024-02-07; First posted 2024-03-06 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Prostate Cancer
Keywords: Transperineal Prostate Biopsy
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Virtual Reality Device (Experimental): The VR device used is the Flowly biofeedback virtual headset. This device uses calming immersive virtual worlds along with breathing exercises and a heart rate monitor to guide patients through meditated breathing exercises. The Flowly app is based on a smartphone which will be purchased through the department and used by all participants. The account used is a generic account for our department. No patient information or individualized accounts will be needed. No patient information or data will be collected.
  Interventions: Other: Virtual Reality Headset; Other: Standard of Care
- Aromatherapy (Experimental): The aromatherapy arm will utilize one standardized patch with a peppermint/lavender scent based on prior research and experience.
  Interventions: Other: Aromatherapy Patch; Other: Standard of Care
- Virtual Reality and Aromatherapy (Experimental): This arm will combine both the Virtual Reality arm and the aromatherapy arm procedure.
  Interventions: Other: Virtual Reality Headset; Other: Aromatherapy Patch; Other: Standard of Care
- Standard of Care (Active Comparator): Participant will undergo transperineal prostate biopsy as standard of care.
  Interventions: Other: Standard of Care

INTERVENTIONS:
Other: Virtual Reality Headset — The interventions are for supportive care ONLY.
  Arms: Virtual Reality Device; Virtual Reality and Aromatherapy
Other: Aromatherapy Patch — The interventions are for supportive care ONLY.
  Arms: Aromatherapy; Virtual Reality and Aromatherapy
Other: Standard of Care — Participant will undergo a transperineal prostate biopsy.

SUMMARY:
The purpose of this study is to evaluate if a VR headset and/or aromatherapy can be used to reduce patient pain, anxiety, and embarrassment during a transperineal biopsy (TPBx) compared to standard of care (SOC). The primary objective is to evaluate differences in self-reported pain, fear, or embarrassment during and after the procedure between the VR Group, Aromatherapy Group, VR+Aromatherapy Group, and the Control group.

DETAILED DESCRIPTION:
This is a single-center, randomized controlled trial comparing the use of a virtual reality (VR) device vs. an aromatherapy patch vs. VR+aromatherapy vs. standard of care as a non-anesthetic pain management tool during a transperineal prostate biopsy (TPBx).

208 patients who express interest in participating in the trial will be consented via Redcap. Patients will be centrally, dynamically randomized in a 1:1:1:1 ratio to one of the treatment groups or control group. There will be no subgroup stratification. The randomization will be predetermined by participant ID number. There will be a sealed envelope prepared and labeled with the participant ID that will contain the information for which treatment group a participant is assigned to. Once a participant is consented and assigned an ID, the envelope will be reopened to reveal which intervention the patient will be assigned to.

All participants will take a survey immediately following the procedure and that will conclude their participation in the study.

ELIGIBILITY:
Inclusion Criteria:

* Patient is 18 years or older
* Patient is male
* Patient is due for a transperineal prostate biopsy
* Patient signed and dated informed consent form on Redcap agreeing to participate in the study

Exclusion Criteria:

* Patient has a known psychiatric or mental illness that would impede use of the VR device or aromatherapy patch
* Patient has severe hearing or vision problems that would impair use of the VR headset (under the physician's discretion)
* Patient has a history of seizures or epilepsy or is on a medication that would lower the threshold for a seizure
* Patient has a history of reactions to noxious odors

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 208 (Estimated)
Dates: Start 2024-05-20 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Levels of pain, fear, and embarrassment that each group experienced before the TPBx measured using a self-reported survey that asks about experience prior to biopsy. The survey will be provided after the procedure. | immediately after the biopsy (up to 30 minutes)
  This outcome will be measured in the survey on a likert scale from least (0) to most (10) fear, anxiety, and embarassment.
Levels of pain, fear, and embarrassment that each group experienced during the TPBx measured using a self-reported survey that asks about experience during the biopsy. The survey will be provided after the procedure. | immediately after the biopsy (up to 30 minutes)
  This outcome will be measured in the survey on a likert scale from least (0) to most (10) fear, anxiety, and embarassment.
Levels of pain, fear, and embarrassment that each group experienced after the TPBx measured using a self-reported survey that asks about experience after to biopsy. The survey will be provided after the procedure. | immediately after the biopsy (up to 30 minutes)
  This outcome will be measured in the survey on a likert scale from least (0) to most (10) fear, anxiety, and embarassment.

SECONDARY OUTCOMES:
Proportion of patients undergoing TPBx who would be interested in using a VR device or aromatherapy patch during the procedure. | during enrollment
  Track number of patients approached and number of patients who sign consent.
Safety and feasibility of using a VR device or aromatherapy patch during TPBx via the proportion of procedures completed successfully with no major complications or prolongations. | during the biopsy procedure (up to 30 minutes)
  Track number of procedures completed successfully with no major complications or prolongations per the investigator's discretion.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Jacobs, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center Shadyside Hospital, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No